CLINICAL TRIAL: NCT05912868
Title: Long-term Results in 174 Patients With a Ventral Hernia in the Midline of the Abdominal Wall After EMILOS (Endoscopic Mini/Less Open Sublay) Repair
Brief Title: Endoscopic Mini/Less Open Sublay(EMILOS) Repair
Acronym: EMILOS
Status: Completed | Type: Observational
Sponsor: Diakonie-Klinikum Stuttgart (Other)
Responsible Party: Sponsor
Other Study IDs: 1/2016
Record Dates: First submitted 2023-02-15; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hernia, Ventral
Keywords: Umbilical hernias-Incisional hernias-EMILOS- .
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ventral hernia repair: Endoscopic Mini/Less Open Repair
  Interventions: Device: Endoscopic Mini/Less Open Sublay Repair

INTERVENTIONS:
Device: Endoscopic Mini/Less Open Sublay Repair — The traditional techniques are open sublay or transabdominal intraperitoneal onlay mesh (IPOM) repair. In order to avoid the risks -large trauma to the abdominal wall with pain and infection, lesion of intraabdominal organs - a new hybrid technique - small skin incision, wide endoscopic dissection of the retrorectus space with implantation of a large mesh - was developed (EMILOS -Endoscopic Mini/Less Open Sublay).

SUMMARY:
Ventral hernias in the midline of the abdominal wall are one of the most frequent diseases in general and visceral surgery worldwide. The optimal operative technique is still in discussion. The traditional techniques are open sublay or transabdominal intraperitoneal onlay mesh (IPOM) repair. In order to avoid the risks -large trauma to the abdominal wall with pain and infection, lesion of intraabdominal organs - a new hybrid technique - small skin incision, wide endoscopic dissection of the retrorectus space with implantation of a large mesh - was developed (EMILOS -Endoscopic Mini/Less Open Sublay).

DETAILED DESCRIPTION:
Long-term results in 174 patients with a ventral hernia of the abdominal wall after EMILOS (Endoscopic Mini/Less Open Sublay) repair.

The worldwide most frequently used surgical techniques to repair ventral abdominal wall hernias are the open sublay operation and the transabdominal IPOM (Intra-Peritoneal Onlay Mesh) technique.

Therefore a special questionnaire was developed to send to the patients to evaluate long-term outcome.

ELIGIBILITY:
Inclusion Criteria

* Patients with clinical diagnosis of primary or secondary hernia in the midline of the abdominal wall
* Defect size must be between 2 and 10 cm in width associated with a weak abdominal wall(rectus diastasis)
* Patient must be suitable for general anesthesia
* Patient must have given informed consent
* Patient must be able to understand the principles of operation
* Patient must agree to be incluuded in a follow-up program and to be documented in Herniamed registry

Exclusion Criteria:

* Patients below 18 years of age
* Patients with a defect size below 2 cm
* Patients presenting with loss of domain
* Patients not be able to tolerate general anesthesia
* Patients presenting with excess skin tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the ambulance of one of the three participating hospitals because of pain or a bulge in the midline of the abdominal wall without previous or after previous abdominal operation
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with Hernia recurrence | three years
  prove of hernia defect and hernia sac by questionaire and clinical investigation
Number of patients with bulging in the midline of abdominal wall | three years
  Bulging without prove of a hernia defect by questionaire and clinical investigation

SECONDARY OUTCOMES:
Number of patients suffering from chronic pain | three years
  Asking by questionaire if the patient has pain at rest and under stress in the region of the scar resp. the former hernia defect measured by numeric analog scale (NAS)
Number of patients complaining about a stiff abdominal wall | three years
  Asking by questionaire if the patient has problems to bend down and/or problems to tie shoestrings
Number of patients being satisfied with operation | Three years
  Asking by questionaire if the patient is satisfied with operation and if he would like to have this operation a second time

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Dr.h.c. Bittner, Principal Investigator — unaffiliated, retirement; Dr. Bärbel Kraft, Study Director — Diakonie-Klinikum Stuttgart; Dr. Jochen Schwarz, Study Director — Hernienzentrum Rottenburg; Dr.Stefan Amann, Study Director — Diakoneo Klinik Neudettelsau
Locations (3):
- Germany (3):
  - Diakonie Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Dr.Stefan Amann, Neuendettelsau
  - Hernia Center, Rottenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz J, Reinpold W, Bittner R. Endoscopic mini/less open sublay technique (EMILOS)-a new technique for ventral hernia repair. Langenbecks Arch Surg. 2017 Feb;402(1):173-180. doi: 10.1007/s00423-016-1522-0. Epub 2016 Oct 20. PMID 27766419
- [Background] Bittner R, Bain K, Bansal VK, Berrevoet F, Bingener-Casey J, Chen D, Chen J, Chowbey P, Dietz UA, de Beaux A, Ferzli G, Fortelny R, Hoffmann H, Iskander M, Ji Z, Jorgensen LN, Khullar R, Kirchhoff P, Kockerling F, Kukleta J, LeBlanc K, Li J, Lomanto D, Mayer F, Meytes V, Misra M, Morales-Conde S, Niebuhr H, Radvinsky D, Ramshaw B, Ranev D, Reinpold W, Sharma A, Schrittwieser R, Stechemesser B, Sutedja B, Tang J, Warren J, Weyhe D, Wiegering A, Woeste G, Yao Q. Update of Guidelines for laparoscopic treatment of ventral and incisional abdominal wall hernias (International Endohernia Society (IEHS)): Part B. Surg Endosc. 2019 Nov;33(11):3511-3549. doi: 10.1007/s00464-019-06908-6. Epub 2019 Jul 10. PMID 31292742
- [Background] Reinpold W, Schroder M, Berger C, Stoltenberg W, Kockerling F. MILOS and EMILOS repair of primary umbilical and epigastric hernias. Hernia. 2019 Oct;23(5):935-944. doi: 10.1007/s10029-019-02056-x. Epub 2019 Sep 30. PMID 31571064
- [Background] Reinpold W, Schroder M, Berger C, Nehls J, Schroder A, Hukauf M, Kockerling F, Bittner R. Mini- or Less-open Sublay Operation (MILOS): A New Minimally Invasive Technique for the Extraperitoneal Mesh Repair of Incisional Hernias. Ann Surg. 2019 Apr;269(4):748-755. doi: 10.1097/SLA.0000000000002661. PMID 29342018
- [Background] Kohler G, Luketina RR, Emmanuel K. Sutured repair of primary small umbilical and epigastric hernias: concomitant rectus diastasis is a significant risk factor for recurrence. World J Surg. 2015 Jan;39(1):121-6; discussion 127.. doi: 10.1007/s00268-014-2765-y. PMID 25217109
- [Background] Kockerling F, Simon T, Adolf D, Kockerling D, Mayer F, Reinpold W, Weyhe D, Bittner R. Laparoscopic IPOM versus open sublay technique for elective incisional hernia repair: a registry-based, propensity score-matched comparison of 9907 patients. Surg Endosc. 2019 Oct;33(10):3361-3369. doi: 10.1007/s00464-018-06629-2. Epub 2019 Jan 2. PMID 30604264
- [Background] Belyansky I, Daes J, Radu VG, Balasubramanian R, Reza Zahiri H, Weltz AS, Sibia US, Park A, Novitsky Y. A novel approach using the enhanced-view totally extraperitoneal (eTEP) technique for laparoscopic retromuscular hernia repair. Surg Endosc. 2018 Mar;32(3):1525-1532. doi: 10.1007/s00464-017-5840-2. Epub 2017 Sep 15. PMID 28916960
- [Background] Kohler G, Fischer I, Kaltenbock R, Schrittwieser R. Minimal Invasive Linea Alba Reconstruction for the Treatment of Umbilical and Epigastric Hernias with Coexisting Rectus Abdominis Diastasis. J Laparoendosc Adv Surg Tech A. 2018 Oct;28(10):1223-1228. doi: 10.1089/lap.2018.0018. Epub 2018 Apr 5. PMID 29620963
- [Background] Reinpold W, Kockerling F, Bittner R, Conze J, Fortelny R, Koch A, Kukleta J, Kuthe A, Lorenz R, Stechemesser B. Classification of Rectus Diastasis-A Proposal by the German Hernia Society (DHG) and the International Endohernia Society (IEHS). Front Surg. 2019 Jan 28;6:1. doi: 10.3389/fsurg.2019.00001. eCollection 2019. PMID 30746364